CLINICAL TRIAL: NCT01096147
Title: Octad Study: Evaluation of the Effectiveness of the Octopolar Lead in Patients With Failed Back Surgery Syndrome With Low Back and/or Leg Pain During a One Year Follow-up Period
Brief Title: Efficacy Study of the Octapolar Lead in Patients With Failed Back Surgery Syndrome (FBSS) With Chronic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rik Buschman, PhD (Industry)
Responsible Party: Sponsor-Investigator, Rik Buschman, PhD, Principal Scientist, Medtronic Neuromodulation Europe
Organization: Medtronic Neuromodulation Europe (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Octad study
Record Dates: First submitted 2010-03-08; First posted 2010-03-30 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-11

CONDITIONS: Failed Back Surgery Syndrome
Keywords: FBSS; chronic pain; leg pain; low back pain; spinal cord stimulation
MeSH Terms: conditions — Failed Back Surgery Syndrome; Chronic Pain; Low Back Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SCS (Active Comparator): patients receiving SCS for chronic leg and/or back pain.
  Interventions: Device: Spinal cord stimulation with eight polar electrode

INTERVENTIONS:
Device: Spinal cord stimulation with eight polar electrode — In SCS a lead is positioned in the epidural space on the dorsal aspect of the spinal cord as to produce electrically induced paraesthesia in the painful area.
  Other Names: Spinal column stimulation

SUMMARY:
Spinal cord stimulation (SCS) has been used for over 40 years to treat neuropathic pain. Various clinical studies have shown a beneficial effect of SCS on pain in patients with Failed Back Surgery Syndrome (FBSS). Since more than 2 years the 8-contact points Octad lead has been used and replaced the 4-contact points Quad lead. Even though it seems that eight electrodes has potential advantage over the four electrodes in case of lead migration or disease progress, no clinical data have been published on the effectiveness of SCS using the octopolar epidural lead. The Octad study intents to assess the effectiveness and technical performance of SCS with the Octad® lead for treatment of chronic pain. This study is not set up as a comparison study between the Octad lead and other SCS leads, such as the Quad lead, because the Octad lead is used in most eligible FBSS patients as the standard of care lead.

The study intends to:

1. evaluate the effectiveness of SCS with the Octad® lead on chronic pain in Failed Back Surgery Syndrome patients after 12 months of treatment.
2. collect safety data for SCS with the Octad® lead in patients with refractory chronic pain.

DETAILED DESCRIPTION:
The use of Spinal Cord Stimulation (SCS) for pain control has already a history of more than 40 years. In SCS, a lead is positioned in the epidural space on the dorsal aspect of the spinal cord so as to produce stimulation induced paraesthesia in the painful area. During the last decades many articles have been published, clearly indicating the effectiveness and safety of SCS with quadripolar leads in the pain management of chronic neuropathic pain, and in particular Failed Back Surgery Syndrome (FBSS). Randomized controlled trials demonstrated that compared with re-operation, SCS provides effective pain relief for at least 3 years and compared with conventional non-surgical neuropathic pain management for at least 2 years.

However, SCS-related complications can occur, that can be divided into surgical complications and hardware complications. The hardware technology has substantially improved over the years. Moreover, electrodes have become smaller in shape and easier to navigate through the epidural space; and finally, internal pulse generators have new programming capabilities and a longer battery life span. All these technological developments led to the application of minimally invasive percutaneous stimulation trials for a variety of patients with chronic neuropathic pain. Turner et al performed a meta-analysis of spinal cord stimulation for failed back surgery syndrome publications and reported hardware complications of 24% lead migration, 7% lead failure and 2% pulse generator failure. While this analysis evaluated studies using older hardware systems, there is first evidence that the rate of these complications is lower currently with new systems. In the recently published PROCESS paper, also using quadripolar electrodes, long term follow-up showed that hardware complications were 14%: lead migration, 3% lead failure and no pulse generator failures.

Generally, patients with radicular pain to the lower extremities respond better to spinal cord stimulation than patients with isolated axial low back pain. However, a few studies have shown that axial low back pain in combination with bilateral leg pain, also respond well to spinal cord stimulation. Both four (e.g. quadripolar Quad lead) and eight (e.g. octapolar Octad® lead) electrodes were shown to be effective in treatment of low back and lower extremity pain, with no apparent advantage of one system over the other. In the recent PROCESS study publication, the reduction of SCS on low-back pain was not-statistically significant when compared to baseline. Even though it seems that eight electrodes may have the potential advantage in case of lead migration or disease progress, no clinical data have been published on the effectiveness of SCS using the octopolar epidural lead. The Octad study is a prospective, multi-center, open-label, non-randomized, interventional study designed to assess the effectiveness and technical performance of SCS with the Octad® lead for treatment of chronic pain. This study is not set up as a comparison study between the Octad lead and other SCS leads, such as the Quad lead, because the Octad lead is used in most eligible FBSS patients as the standard of care lead.

ELIGIBILITY:
Inclusion Criteria:

1. FBSS patients with neuropathic pain in low-back and/or legs who have not reached their therapy goal with other treatment interventions
2. ≥ 18 years of age
3. Chronic pain as a result of FBSS that exists for at least 6 months
4. Mean pain intensity in the legs should be 5 or higher measured on Visual Analogue Scale (VAS).
5. Patient has been informed of the study procedures and has given written informed consent.
6. Patient willing to comply with study protocol including attending the study visits.

Exclusion Criteria:

1. Expected inability of patients to receive or properly operate the spinal cord stimulation system
2. History of coagulation disorders, lupus erythematosus, diabetic neuropathy, rheumatoid arthritis or morbus Bechterew
3. Active malignancy
4. Addiction to any of the following: drugs, alcohol (5E/day) and/or medication
5. Evidence of an active disruptive psychiatric disorder or other known condition significant enough to impact perception of pain, compliance to intervention and/or ability to evaluate treatment outcome as determined by investigator
6. Immune deficiency (HIV positive, immunosuppressive, etc.)
7. Life expectancy < 1 year
8. Local infection or other skin disorder at site of incision
9. Pregnancy
10. Other implanted active medical device
11. Participation in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-02; Primary Completion 2013-03 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pain suppression in low back and/or leg | 12 months
  Evaluate the evolution of pain control with the octopolar Octad® lead assessed by a decrease in VAS for leg (and low-back pain separately, if applicable) during 12 months follow-up. Actual pain, the least pain during the last week and the worst pain during the last week are scored.

SECONDARY OUTCOMES:
adverse events related to SCS | 12 months
  Clinical (such as surgery related infections) and technical (such as lead fractures) adverse events will be collected continuously in all patients during a period of 12 months post implant.
quality of life | 12 months
  Quality of life assessed by EuroQol group - 5 Dimensions (EQ-5D)
sleep | 12 months
  Sleep is assessed by a 3 item questionnaire on sleep quality, falling asleep and waking up from pain.
pain medication intake | 12 months
  Data will be collected at specific times on health service resourse use of concomitant pain medication such as opioids.
Healthcare resource utilization | 12 months
  Data will be collected at specific times on health service resourse use of concomitant non-drug therapy use, such as physiotherapy, related to FBSS.
preferred stimulation settings | 12 months
  Characterization of pulsegenerator parameters, such as amplitude, pulse width, stimulation frequency, electrode configuration (positive and negative poles), number of stimulation programs, and stimulation duration is done at specific times.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Ver Donck, MD PhD, Principal Investigator — Hospital St Jan, Brugge, Belgium; Kliment P Gatzinsky, MD PhD, Principal Investigator — Sahlgrenska University Hospital; Roald Baardsen, MD PhD, Principal Investigator — University hospital Stavanger, Stavanger, Norway
Locations (8):
- Belgium (6):
  - Hospital ZNA Middelheim, Antwerp
  - Hospital St Jan, Bruges
  - Hospital Alma Eeklo, Eeklo
  - University Hospital Gent, Ghent
  - Hospital Nicolaas, Sint-Niklaas
  - St Elisabeth, Zottegem
- Stavanger University Hospital, Stavanger, Norway
- Shalgrenska Hospital, Gothenburg, Sweden